CLINICAL TRIAL: NCT00767065
Title: The Role of Early X-Ray Cardiac Computed Tomography in Patients Admitted With Acute Chest Pain
Brief Title: Early Cardiac Computed Tomography (CT) In Patients Admitted With Acute Chest Pain
Acronym: EXACCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); British Heart Foundation (Other)
Responsible Party: Dr Simon Padley, Chelsea and Westminster NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CWRT/SP2008/1
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-09

CONDITIONS: Acute Chest Pain
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiac Computed Tomography (CCT) (Active Comparator): Patients randomised to the CCT arm will undergo 128-channel cardiac computed tomography with delayed acquisition. CCT will be available Monday to Friday from 9am until 5pm. Patients will be entered into the study provided CCT can be undertaken within 24 hours of troponin result. Therefore, the only period during which a patient will be ineligible for inclusion will be between 5pm on a Friday and 9am the following Sunday. Studies will be reported at CWH by one of 2 experienced radiologists trained in CCT and results passed to the referring team on the same day.
  Interventions: Radiation: Cardiac Computed Tomography
- Standard Care Arm (Active Comparator): Patients randomised to the standard care arm will undergo further care as dictated by the responsible clinician. Except for CCT, all standard investigations will be available to the responsible clinician and may be used at their discretion. CCT does not form part of current in-patient management at our hospital.
  Interventions: Other: Standard care

INTERVENTIONS:
Radiation: Cardiac Computed Tomography — Patients randomised to the CCT arm will undergo 128-channel cardiac computed tomography with delayed acquisition. Patients will receive beta-blockade if necessary prior to the scan to achieve a heart rate of less than 70/min. An unenhanced scan will be performed in all patients to assess coronary artery calcium score. Patients will then undergo contrast enhanced CCT. After a bolus tracking acquisition, injection of 120mls iodinated contrast at 5ml/s will be followed by 40ml normal saline/contrast (in 50:50 proportion), also at 5ml/s. Imaging will be performed with a gated cardiac CT protocol. Where possible (stable rhythm and heart rate <70bpm) a low dose technique will be utilised. When not possible a retrospective gating method will be employed. In the latter case the ECG will be used to assign the images to their respective phases of the cardiac cycle. 10 minutes after contrast injection, a second prospectively gated scan will be acquired to assess myocardial enhancement patterns.
  Arms: Cardiac Computed Tomography (CCT)
Other: Standard care — Further investigations as decided by the patient's clinical team, according to best normal practice. These may include some or all of: further blood tests, exercise stress testing and myocardial perfusion scintigraphy. These may be conducted either during the initial hospital admission, or subsequently as an outpatient.
  Arms: Standard Care Arm

SUMMARY:
This is a randomised trial comparing early Cardiac Computed Tomography (CCT) to current standard practice for diagnosis of acute chest pain in patients at low to intermediate risk of having coronary artery disease (CAD), in a UK setting. We hypothesise that early CCT can reduce length of admission, reduce NHS costs and improve quality of life whilst being at least as safe as standard practice.

DETAILED DESCRIPTION:
Coronary Artery Disease (CAD) kills more people in the UK than any other condition, and causes symptoms of angina (chest pain) in many more. Acute chest pain accounts for approximately 600,000 NHS admissions per annum, but this includes many other types of chest pain not due to heart problems. Examination, blood tests and an electrocardiogram (ECG) are used to try and decide the cause of chest pain.

Many patients have a low risk of CAD and can be discharged without further investigation. Others are at high risk of CAD and must have further tests such as invasive coronary angiography. Unfortunately in many patients the initial tests are equivocal and they are felt to have an intermediate probability of CAD. Investigation of symptoms in this group may take place in the in-patient setting, warranting a hospital stay of several days, or alternatively some investigations may be performed as an out-patient with subsequent time spent on waiting lists. This results in extensive use of NHS resources and anxiety for the patients whilst awaiting diagnosis, often needlessly as approximately half of patients admitted with acute chest pain are eventually discharged without a cardiac cause found.

The new technique of cardiac computed tomography (CCT) offers rapid non-invasive diagnosis of CAD. If disease is detected further investigations can be planned; when excluded, patients may be safely discharged. Detection of clinically insignificant disease will initiate primary preventative strategies but excludes CAD as the cause of acute symptoms. We will randomise 250 patients presenting to Chelsea and Westminster Hospital with acute chest pain who have intermediate likelihood of CAD to early CCT or current standard practice. We hypothesise that, when compared to standard practice, early CCT will reduce admission length, reduce NHS and other costs and improve quality of life without an increase in adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Admission with suspected cardiac chest pain
2. >40 years of age
3. EITHER Low likelihood of CAD according to DFC and troponin>0.03 but <3 OR Intermediate likelihood of CAD according to DFC
4. Written informed consent

Exclusion Criteria:

1. ECG consistent with acute myocardial infarction (ST elevation, new left bundle branch block)
2. Ongoing chest pain with dynamic ECG changes
3. Haemodynamic or respiratory instability
4. Serum troponin ≥3
5. Previous percutaneous coronary intervention or coronary artery bypass grafting
6. Admission to hospital between 5pm Friday and 9am Sunday
7. Contraindication to negative chronotropic agents
8. Maximum heart rate >70bpm (including after pharmacologic treatment)
9. Renal dysfunction (Creat>150 micromol/l)
10. Pregnancy or childbearing potential
11. Allergy or previous intolerance of iodinated contrast

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Length of hospital admission | At the end of initial hospital admission

SECONDARY OUTCOMES:
NHS costs and cost-effectiveness over a one-year period | One year
Patient quality of life at 1, 6 and 12 months after admission | 1 year
Patient anxiety about symptoms 1, 6 and 12 months after admission | 1 year
The incidence of major adverse cardiovascular events (MACE) over a one year period. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Simon Padley, MB BS BSc FRCP FRCR, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom